CLINICAL TRIAL: NCT02267889
Title: A Pilot Study on the Role pf Ganglionated Plexus Ablation for Catheter Ablation of Atrial Fibrillation.
Brief Title: Ganglionated Plexus Ablation For Treatment of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spectrum Dynamics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDRBH01
Record Dates: First submitted 2014-10-14; First posted 2014-10-20 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Atrial Fibrillation
Keywords: Ganglionated plexi
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Image guided GP ablation (Experimental): Use of cardiac nuclear imaging data to guide GP ablation procedures.
  Interventions: Procedure: Image guided GP ablation; Device: D-SPECT dedicated cardiac nuclear camera

INTERVENTIONS:
Procedure: Image guided GP ablation — 3D imaging data from the D-SPECT system will be used to visualise the GP and guide the location of catheter ablation sites during the electrophysiology procedure.
  Other Names: D-SPECT dedicated cardiac nuclear camera
Device: D-SPECT dedicated cardiac nuclear camera

SUMMARY:
This study evaluates the effect of catheter ablation of ganglionated plexi (GP) for the treatment of adult patients with atrial fibrillation heart arrhythmias. The location of GP will be demonstrated by a novel nuclear imaging cardiac camera. 3D images from the cardiac camera will guide the GP ablation procedure.

DETAILED DESCRIPTION:
Catheter ablation procedures are nowadays routine procedures in patients with drug-refractory atrial fibrillation (AF). However, ablation success for patients even in the early stages of AF is currently only around 70% and may require multiple procedures.

The intrinsic cardiac autonomic nervous system (ANS), which forms a neural network, has been shown to be a critical element responsible for the initiation and maintenance of AF. Autonomic inputs to the heart converge at several locations; these convergence points are typically embedded in the epicardial fat pads and form ganglionated plexi (GP) that contain autonomic ganglia and nerves. In human hearts, there are at least 7 GP and the 4 major left atrial GP are located around the antrum of the pulmonary veins (PVs). High-frequency stimulation (HFS; 20 Hz, 10-150 V and pulse width 1-10 ms) can localize GP during an invasive electrophysiology (EP) study.

A novel dedicated cardiac nuclear imaging camera with solid-state detectors (D-SPECT, Spectrum Dynamics) has demonstrated significantly improved sensitivity and image resolution and can provide novel imaging information on previously 'invisible' structures like the GP. Using this 3D image information to guide GP ablation could significantly facilitate AF ablation and result in improved ablation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal or early persistent atrial fibrillation with ongoing AF for less than 1 week
* Able to give written informed consent
* Age >18 years old and ≤ 80 years
* Fulfil established clinical criteria for catheter ablation of atrial fibrillation
* Normal left ventricular (LV) ejection fraction and no evidence of significant structural heart disease

Exclusion Criteria:

* Reversible cause of atrial fibrillation
* Recent cardiovascular event including transient ischaemic attack (TIA)
* Intolerance or unwillingness to oral anticoagulation with Warfarin
* Bleeding disorder
* Contraindication to computed tomography (CT) scan
* Presence of intracardiac thrombus
* Vascular disorder preventing access to femoral veins
* Cardiac congenital abnormality
* Severe, life threatening non cardiac disease
* Active malignant disease or recent (<5 years) malignant disease
* Presence of atrial septal defect (ASD) or patent foramen ovale (PFO) closure device
* Unable or unwilling to comply with follow-up requirements
* Patients on amiodarone until less than 3 months prior to the screening visit
* Left atrium size > 5.5 cm on parasternal diameter in transthoracic echocardiography (TTE)
* Renal impairment
* Pregnancy

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Termination of atrial fibrillation during image guided ablation | At the time of the ablation procedure.
Freedom from atrial fibrillation/flutter/tachycardia (>30 seconds) off antiarrhythmic medication at the end of 12 months following the index ablation procedure. | 12 months post the index ablation procedure.

SECONDARY OUTCOMES:
Time to first recurrence of atrial fibrillation/flutter/tachycardia (>30 seconds) | Up to 12 months from the index ablation procedure
Freedom from atrial fibrillation on previously failed antiarrhythmic medication | 12 months from the index ablation procedure.
Atrial fibrillation/flutter/tachycardia (>30 seconds) burden at 12 months post the index ablation procedure. | 12 months from the index ablation procedure.
  AF/flutter/tachycardia burden will be modelled as a continuous variable with the number of episodes recorded.
Left atrial transport function | 6 months and 12 months post the index ablation procedure
  Left atrial transport function will be assessed by echo as a categorical variable with 3 categories; poor, moderately impaired and normal.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Ernst, MD, Principal Investigator — The Royal Brompton Hospital, London, UK
Locations (1):
- The Royal Brompton Hospital, London, United Kingdom